CLINICAL TRIAL: NCT01613872
Title: The Effects of Mindfulness Based Stress Reduction on Patients With Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Ross D. Zafonte, MD, Chair, Physical Medicine and Rehabilitation, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-P-000557/1
Record Dates: First submitted 2012-05-29; First posted 2012-06-07 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Traumatic Brain Injury; Brain Injury; Stress
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Wait List Control
- Mindfulness Based Stress Reduction (Experimental): An 8 week standardized protocol of stress reduction using gentle yoga and meditation
  Interventions: Other: Mindfulness Based Stress Reduction

INTERVENTIONS:
Other: Mindfulness Based Stress Reduction — An 8 week protocol of stress reduction sessions using gentle yoga and breath meditation
  Arms: Mindfulness Based Stress Reduction

SUMMARY:
This study is studying the effects of Mindfulness Based Stress Reduction (MBSR), a standard protocol of gentle yoga and breath meditation, on patients with Traumatic Brain Injury (TBI). The investigators are testing whether this intervention can help improve the stress response and increase resiliency and mindfulness for patients with TBI, which may lead to improved symptoms and neurocognitive function.

ELIGIBILITY:
Inclusion Criteria:

* TBI > 1 year prior to enrollment
* Ages 30-50
* Right handed participants
* History of acute inpatient rehabilitation stay of ≥ 1 night

Exclusion Criteria:

* Non-English speaking (because this is a group intervention, it requires a common language)
* Dependent with activities of daily living (ADLs)
* Phone screen (TICS-1) > 30
* Rivermead Post-Concussion Questionnaire Score < 21
* Actively practicing meditation and/or yoga or have taken a meditation/yoga class in the last 12 months
* Signs or symptoms of upper motor neuron syndrome
* Any major major systemic illness or unstable condition which could interfere with protocol compliance, including the diagnosis of major depression
* Active psychiatric disease that would interfere with participation in the trial
* Psychotic features, agitation, or behavioral problems within the last 3 months
* History of alcohol/substance abuse or dependence within the past 2 years
* Neurosurgical intervention affecting brain parenchyma
* Reported sequelae from brain lesions or head trauma prior to most recent brain injury
* Seizure activity or treatment for seizures
* Use of investigational agents
* Participating in other clinical studies involving neuropsychological measures collected more than one time per year
* Any involvement in legal matters (workers' compensation, litigation, et al), past, present, or anticipated in the future, related to the TBI
* Unable to undergo MRI for any reason such as claustrophobia, presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Feasibility and Safety | 8 weeks
  Benchmark measurements of attendance, home practice, adverse events, and focused interviews

SECONDARY OUTCOMES:
Neuropsychological Testing | 8 weeks
  A neuropsychological battery to be assessed at baseline and post-intervention.
Advanced MRI | 8 weeks
  Advanced MRI will be used to assess any potential changes (neuroplasticity)
Questionnaires | 8 weeks
  Questionnaires to assess subjective experiences with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ross Zafonte, DO, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States